CLINICAL TRIAL: NCT02740855
Title: Endtidal Ethanol in Sclerotherapy
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Endtidal ethanol
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Ethanol Concentration
Keywords: sclerotherapy; ethanol; pulmonal hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Device: Alcomed 3011® — Endtidal ethanol measurement

SUMMARY:
During the ethanol sclerotherapy procedure, the investigators will record doses of and time of ethanol injections and record ethanol concentrations in endtidal breath every 5 minutes. Furthermore after every ethanol injection the concentration will be measured every minute for 5 minutes. To do so, the investigators will attach a breath alcohol testing device to the expiratory carbon dioxide measuring unit. Since this is the new standard of the university hospital Berne all patients undergo the same procedure. There is no study specific intervention. In this study the investigators will only document the breath alcohol levels, doses and timing of ethanol injections. All other data will be obtained from the anesthesia information system. During the two months of the study, the investigators will also record endtidal ethanol concentration after anesthesia in the postoperative care unit discharge from the unit.

The intention is to show the correlation between injected ethanol doses and measured endtidal ethanol concentration over the entire time of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* undergoing ethanol sclerotherapy at the university hospital Berne

Exclusion Criteria:

* under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing ethanol sclerotherapy at the university hospital Berne over the age of 18.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Endtidal ethanol concentrations in mg/dl over time | 1 year 2 months

SECONDARY OUTCOMES:
Bloodpressure in mmHg over time | 1 year 2 months
Bloodpressure in mmHg over injected peripheral ethanol volume | 1 year 2 months
Pulse rate in beats er minute over time | 1 year 2 months
Pulse rate in beats er minute over injected peripheral ethanol volume | 1 year 2 months
Endtidal ethanol concentrations in mg/dl over injected ethanol volume | 1 year 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland